CLINICAL TRIAL: NCT00500552
Title: Metabolic Alteration With Perhexiline Therapy in Patients With Hypertrophic Cardiomyopathy (METAL-HCM Study)
Brief Title: Perhexiline Therapy in Patients With Hypertrophic Cardiomyopathy
Acronym: METAL-HCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Birmingham (Other)
Collaborators: British Heart Foundation (Other); University College London Hospitals (Other); University of Oxford (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRK 2848, 05/Q2707/325; PG/05/087
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-08

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Perhexiline; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Perhexiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Perhexiline/Placebo

SUMMARY:
Hypertrophic Cardiomyopathy (HCM) is a relatively common inherited heart muscle disease. Many patients experience symptoms of breathlessness, fatigue and chest pain. These symptoms are not always controlled with current therapies.

Recently the investigators showed that a drug called Perhexiline markedly improved exercise capacity and symptoms in patients with heart failure. In this proposal the investigators wish to test whether Perhexiline improves exercise capacity and relieves symptoms in patients with HCM

DETAILED DESCRIPTION:
Background:

Hypertrophic cardiomyopathy (HCM) is a complex and relatively common genetic cardiac disease and it is the most common cause of sudden cardiac death in young people, including trained athletes. In a recent study using in vivo cardiac MR spectroscopy resting PCr/ATP ratio was diminished in patients with sarcomeric HCM, indicating reduced energy availability. Importantly patients with genotypic HCM who did not yet have hypertrophy had a similar degree of impairment of cardiac PCr/ATP ratio as do patients with marked hypertrophy, implying that the disturbance may be an early feature of the disease and is not simply due to the hypertrophy. In medically refractory patients with obstruction, surgical myectomy or alcohol septal ablation may be very effective. However in patients with non obstructive HCM with symptoms refractory to standard drug therapy, there are no therapeutic options (apart from cardiac transplant in very severe cases). Recently, our group showed that Perhexiline, an antianginal agent with an oxygen-sparing metabolic effect which increases the efficiency of energy production by shifting substrate utilisation from free fatty acids towards glucose, was highly effective in improving symptoms, exercise capacity (Vo2max) and cardiac function in patients with systolic heart failure of both ischaemic and non ischaemic aetiology.

Hypothesis:

The investigators postulate that Perhexiline will improve symptomatic status, peak oxygen consumption, resting and exercise diastolic function and that this will be associated with improvement in myocardial energetic status in highly symptomatic medically refractory patients with non obstructive HCM.

Methods and design:

The study is a multi-centre randomised double blind placebo controlled trial. 50 patients who meet the entry criteria and provide written informed consent will be recruited to the study. Patients will be recruited from cardiomyopathy clinics in London, Birmingham and Oxford.

The primary end point will be peak oxygen consumption (Vo2max). Secondary end points will be resting myocardial energetics (31P Cardiac MR Spectroscopy), resting and exercise diastolic function (Myocardial Nuclear studies), Symptomatic Status (Minnesota questionnaire)and LV function (Speckle Tracking Echo measurements).

After the investigations have been performed, subjects will be randomised to receive either 100 mg of Perhexiline a day or placebo for 3 months. Following completions of three months therapy, these investigations will be repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic Hypertrophic Cardiomyopathy patients
2. Abnormal Peak VO2
3. No significant LVOT obstruction at rest (gradient < 30mmHg)
4. Sinus rhythm

Exclusion Criteria:

1. Abnormal LFT.
2. Concomitant use of amiodarone
3. Pre-existing evidence of peripheral neuropathy.
4. Women of childbearing potential.
5. Patients with ICD's will be excluded from the MR part of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption (Vo2max) | 3-4 months

SECONDARY OUTCOMES:
LV function (TDI and 2DS Echo) | 3-4 months
Symptomatic Status (questionnaire) | 3-4 months
Resting myocardial energetics (31P Cardiac MR Spectroscopy) | 3-4 months
Diastolic function at rest and during exercise (Nuclear studies) | 3-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frenneaux, MD, Principal Investigator — University of Birmingham
Locations (3):
- United Kingdom (3):
  - heart Hospital, University College of London NHS, London, London
  - University of Birmingham, Birmingham, West Midlands
  - University of Oxford, Oxford

REFERENCES:
- [Derived] Abozguia K, Elliott P, McKenna W, Phan TT, Nallur-Shivu G, Ahmed I, Maher AR, Kaur K, Taylor J, Henning A, Ashrafian H, Watkins H, Frenneaux M. Metabolic modulator perhexiline corrects energy deficiency and improves exercise capacity in symptomatic hypertrophic cardiomyopathy. Circulation. 2010 Oct 19;122(16):1562-9. doi: 10.1161/CIRCULATIONAHA.109.934059. Epub 2010 Oct 4. PMID 20921440